CLINICAL TRIAL: NCT00137124
Title: Transport and Metabolism of L-arginine: Role for Endothelial Dysfunction in Essential Hypertension
Brief Title: L-Arginine Metabolism in Essential Hypertension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KFO 106 TP8
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: L-Arginine — oral administration of L-arginine for 4 weeks

SUMMARY:
Essential hypertension is characterized by impaired endothelial function. Data derived from normotensive subjects with a genetic predisposition to arterial hypertension suggest that endothelial dysfunction is a cause rather than a consequence of the condition. Given that, in normotensive offspring of hypertensive parents, impaired endothelium dependent vasodilation can be restored by supplementation of the nitric oxide (NO) precursor L-arginine, a defect in the L-arginine/NO pathway can be postulated. The investigators at the University of Erlangen-Nuremberg, hypothesize that impaired endothelial function in essential hypertension is associated with alterations in L-arginine metabolism and transport. This study will determine whether metabolism and transport of L-arginine are altered in patients with essential hypertension and whether these potential alterations can be targeted therapeutically.

ELIGIBILITY:
Inclusion Criteria:

* Males, ages 18-65
* Male and female healthy control subjects ages 18-65

Exclusion Criteria:

* Any other coexisting condition
* Advanced damage of vital organs (grade III und IV retinopathy)
* Therapy with a not approved concomitant medication in the last 4 weeks prior to intake of the first trial medication, especially lipid lowering and antidiabetic medications (washout phase)
* Blood donation within the last 4 weeks
* Patients with arterial fibrillation or atrioventricular (AV)-block (II and more)
* Patients with anamnestic myocardial infarct
* Patients with depression
* Patients with seizure disorders
* Patients with unstable angina pectoris including electrocardiogram (ECG)-aberrations or cardiac insufficiency New York Heart Association (NYHA) Stadium III and IV
* History of a malignant illness with the exception of those patients who have recovered for more than 10 years or have a basalioma of the skin.
* Actual or anamnestic alcohol or drug abuse
* History of organ transplant
* Anaphylaxis or known therapy resistance to any of the used test matters.
* Therapy with a not approved concomitant therapy
* Participation in another study within three months prior to study inclusion
* Illnesses, which can influence the pharmacodynamics or pharmacokinetics of the test substance
* Liver or kidney diseases: SGOT, GPT , γ-GT, AP, bilirubin and creatinine above 200% of standard
* Patients who are not sufficiently compliant; or patients who are not capable or willing to appear for controlling visits.
* Severe or unstable medical or psychiatric illnesses, which will, in the estimation of the examiner, endanger the safety of the proband or the successful participation in the study
* Presumed risk of transmission of HIV or hepatitis via blood from the proband

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
meaning of L-arginine transport and metabolism on endothelial function | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Markus P Schlaich, MD, Principal Investigator — CRC, Medizinische Klinik 4 - Nephrology and Hypertension
Locations (1):
- CRC, Medizinische Klinik 4 - Nephrology and Hypertension, University of Erlangen-Nürnberg, Erlangen, Germany